CLINICAL TRIAL: NCT01843296
Title: Comparison of the Effects of Three Methods of Intrathecal Bupivacaine; Bupivacaine-Fentanyl and Bupivacaine-Fentanyl-Magnesium Sulfate on Sensory-Motor Blocks and Postoperative Pain in Patients Undergoing Lumbar Disk Herniation Surgery
Brief Title: Effects of Addition of Magnesium Sulfate in Spinal Anesthesia on Sensory-Motor Blocks and Postoperative Pain in Lumbar Disk Herniation Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Isfahan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Fereidoun Mortazavi Najafabadi, MD, fellowship of neuroanesthesia, Isfahan University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 392022
Record Dates: First submitted 2013-04-24; First posted 2013-04-30 (Estimated); Last update posted 2013-07-02 (Estimated); Status verified 2013-06

CONDITIONS: Lumbar Spine Disc Herniation
Keywords: Spinal Anesthesia; Bupivacaine; Fentanyl; Magnesium sulfate; Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Magnesium Sulfate; Anesthesia, Spinal; Bupivacaine; Fentanyl

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Magnesium (Active Comparator): Patients in group C received a premixed solution of 15 mg hyperbaric bupivacaine 0.5% (3 ml) and 25 µg fentanyl (0.5cc) and 50 mg of magnesium sulfate 50% (0.1 ml) (Pasteur Institute Co, Tehran, Iran) for spinal anesthesia
  Interventions: Drug: Magnesium Sulfate; Procedure: Spinal Anesthesia; Drug: Bupivacaine; Drug: Fentanyl
- Fentanyl (Active Comparator): Patients in Fentanyl group received a premixed solution of of 15 mg hyperbaric bupivacaine 0.5% (3 ml) and 25 µg fentanyl (0.5cc),plus 0.1 cc preservative free 0.9% normal saline for spinal anesthesia
  Interventions: Procedure: Spinal Anesthesia; Drug: Bupivacaine; Drug: Fentanyl
- Bupivacaine (Active Comparator): Patients in Bupivacaine group(control) received a premixed solution of 15 mg of hyperbaric bupivacaine 0.5% (3 ml), plus 0.6 cc preservative free 0.9% normal saline for spinal anesthesia
  Interventions: Procedure: Spinal Anesthesia; Drug: Bupivacaine

INTERVENTIONS:
Drug: Magnesium Sulfate — Injection of 50 mg of magnesium sulfate 50% (0.1 ml),intrathecally.
  Other Names: Magnesium sulfate 50%
  Arms: Magnesium
Procedure: Spinal Anesthesia — Lumbar puncture was performed in sitting position,at the one level above iliac crest. Using a median approach, a 25-G Quincke needle was introduced with the needle aperture directed laterally.
Drug: Bupivacaine
  Other Names: Marcaine
Drug: Fentanyl
  Other Names: Sublimaze
  Arms: Fentanyl; Magnesium

SUMMARY:
The purpose of this study is to Compare three methods of intrathecal bupivacaine; bupivacaine-fentanyl; bupivacaine-fentanyl-magnesium sulfate on sensory-motor blocks and postoperative pain in patients undergoing lumbar disk herniation surgery.

DETAILED DESCRIPTION:
* Comparison three methods of intrathecal bupivacaine;bupivacaine-fentanyl;bupivacaine-fentanyl-magnesium sulfate on sensory-motor blocks in patients undergoing lumbar disk herniation surgery
* Comparison three methods of intrathecal bupivacaine;bupivacaine-fentanyl;bupivacaine-fentanyl-magnesium sulfate on postoperative pain in patients undergoing lumbar disk herniation surgery
* Comparison three methods of intrathecal bupivacaine;bupivacaine-fentanyl;bupivacaine-fentanyl-magnesium sulfate on postoperative side effects in patients undergoing lumbar disk herniation surgery

ELIGIBILITY:
Inclusion Criteria:

* Candidate for lumbar disk herniation surgery
* No contraindication to the spinal anesthesia
* No history of allergy to opioids and magnesium sulfate
* No peripheral or central neuropathies
* No previous history of surgery on same disk level

Exclusion Criteria:

* Patients with intraoperative tearing of dural suc
* Occuring of inadvertent intraoperative complications such as bleeding

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2012-11; Primary Completion 2012-12 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
The onset of sensory block | From intrathecal injection until the onset of sensory block assessed up to 15 minutes
  Comparing the onset of sensory blocks to T10 (10th thoracic dermatome) assessed by pinprick test.
The complete motor block | From intrathecal injection until the onset of complete motor block assessed up to 15 minutes
  Time to complete motor block after intrathecal injection as assess using a modified Bromage scale
The sensory block regression | From intrathecal injection until the sensory block reression to (T10) assessed up to 6 hours
  The sensory block regression to (T10) dermatome
The full motor recovery | From intrathecal injection until the full motor recovery assessed up to 6 hours
  Full motor recovery was defined as zero on the Bromage scale.
The Pain Score | The first 24 hours after spinal anesthesia
  Using VAS (Visual Analogue Score) system
Time to first analgesic requirement | During first 24 hours after spinal anesthesia
  Time to first analgesic requirement was measured from the time of spinal injection to the first time at which the patient complained of pain in the postoperative period

SECONDARY OUTCOMES:
Mean Arterial Blood Pressure | First hour after spinal anesthesia
  To compare blood pressure alteration and hypotension between three groups
Heart Rate | First hour after spinal anesthesia
  To compare heart rate variation and bradycardia between three groups

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Ali Attari, MD, Study Chair — Isfahan University of Medical Sciences
Locations (1):
- Alzahra, Isfahan, Isfahan, Iran